CLINICAL TRIAL: NCT07183410
Title: Impact of Blood Cultures Drawn From Arterial Lines on the Incidence of Contamination, Detection of Bacteremia, and Blood Culture Volume: an Observational Study
Brief Title: Impact of Blood Cultures Drawn From Arterial Lines on the Incidence of Contamination, Detection of Bacteremia, and Blood Culture Volume
Status: Not yet recruiting | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, sara dichtwald, Dr, Meir Medical Center
Other Study IDs: MMC-0234-25-
Record Dates: First submitted 2025-09-14; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Bacteremia
MeSH Terms: conditions — Bacteremia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cultures from arterial line: From each patient enrolled in the study, two sets of blood cultures will be drawn: one set (2 bottles) from an arterial line and one set from peripheral venous puncture. Each patient will be both the study and the control group for himself: The comparison will be between the arterial line vs. the peripheral vein puncture set.
  In addition, we will also perform a before and after intervention analysis- to examine whether the implementation of the new protocol improved the rate of appropriate blood culture volume and number of culture drawn from the patient .
  Interventions: Diagnostic Test: Blood culture taken from an arterial catheter
- Cultures from peripheral venous puncture: From each patient enrolled in the study, two sets of blood cultures will be drawn: one set (2 bottles) from an arterial line and one set from peripheral venous puncture. Each patient will be both the study and the control group for himself: The comparison will be between the arterial line vs. the peripheral vein puncture set.
  In addition, we will also perform a before and after intervention analysis- to examine whether the implementation of the new protocol improved the rate of appropriate blood culture volume and number of culture drawn from the patient .

INTERVENTIONS:
Diagnostic Test: Blood culture taken from an arterial catheter — Blood culture taken from an arterial catheter (instead of peripheral venous puncture)
  Groups: Cultures from arterial line

SUMMARY:
Taking blood cultures is an important and very common procedure in intensive care units due to the high incidence of sepsis and the need for rapid and accurate identification of bacteremia. However, despite the importance of taking a sufficient volume of blood for the purpose of identifying bacterial growth in the blood, the average blood volume in blood cultures at our institution ranges from 3.5-4 ml per bottle (where the desired volume is 10 ml). Taking an insufficient amount of blood reduces the ability of the bacteriological laboratory to detect bacterial growth and thus may lead to a delay or missed diagnosis of bacteremia, identification of the pathogen, and adjustment of appropriate treatment according to sensitivities.

In intensive care units, most patients are monitored using an arterial catheter, which allows for frequent blood tests without the need to puncture the patient. Following recently published studies that showed that there is no significant difference in the incidence of contamination when taking blood cultures from an arterial catheter compared to a peripheral vein puncture, and in order to improve our ability to identify bacteremia, it was decided to implement a new protocol in the General Intensive Care Unit that includes taking blood cultures from an arterial catheter. According to the new protocol, it was decided that when taking blood cultures from a patient with an arterial catheter, one pair of cultures should be taken from the arterial catheter and another pair from a peripheral vein puncture.

In this study, we would like to examine the contamination rate of blood cultures, the identification of true bacteremia, and the collection of appropriate blood volume and number of blood specimens taken in patients hospitalized in the General Intensive Care Unit at our institution, while analyzing differences between the period before the implementation of the new protocol and the period after the implementation, and differences between cultures taken from an arterial catheter and from a peripheral vein puncture.

ELIGIBILITY:
Inclusion Criteria:All patients aged 18-99 years who had blood cultures taken as part of their routine care in the intensive care unit for any reason, from January 2024 to January 2027.

-

Exclusion Criteria:Missing data or patients who did not fullfil the above criteria.

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the intensive care unit in our hospital between January 2024 and January 2027 who had blood cultures taken as part of their routine care.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Contamination and real bacteremia detection rates | One week following blood cultures collection
  To examine whether there are differences between the contamination rate and the detection rate of true bacteremia between blood cultures from an arterial catheter and blood cultures from a fresh puncture of a peripheral vein.

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel